CLINICAL TRIAL: NCT02884622
Title: DNA Methylation and Lung Disease in Cystic Fibrosis
Acronym: METHYLCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Vaincre la Mucoviscidose (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9133
Record Dates: First submitted 2016-08-16; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2013-03

CONDITIONS: Cystic Fibrosis
Keywords: Lung disease; Epigenetics; DNA methylation; Modifier genes
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CF patients (Other): CF patients with the same procedures as in the usual management of routine care, only the sampling nasal epithelial cells will be added and blood sampling will be collected for this study
  Interventions: Other: nasal epithelial; Other: Blood sampling

INTERVENTIONS:
Other: nasal epithelial — CF patients with the same procedures as in the usual management of routine care, only the sampling nasal epithelial cells will be added
Other: Blood sampling — CF patients with the same procedures as in the usual management of routine care, only the sampling 5ml additional blood will be taken

SUMMARY:
Lung disease progression is variable among cystic fibrosis (CF) patients and depends on DNA mutations in the CFTR gene, polymorphic variations in disease-modifier genes and environmental exposure. The contribution of genetic factors has been extensively investigated, whereas the mechanism whereby environmental factors modulate the lung disease is unknown. Because these factors can affect the epigenome, investigators hypothesized that DNA methylation variations at disease-modifier genes modulate the lung function in CF patients.

DETAILED DESCRIPTION:
Lung disease progression is variable among cystic fibrosis (CF) patients and depends on DNA mutations in the CFTR gene, polymorphic variations in disease-modifier genes and environmental exposure. The contribution of genetic factors has been extensively investigated, whereas the mechanism whereby environmental factors modulate the lung disease is unknown. Because these factors can affect the epigenome, investigators hypothesized that DNA methylation variations at disease-modifier genes modulate the lung function in CF patients.

The investigators analyzed DNA methylation levels in the promoter of fourteen lung disease-modifier genes and showed that DNA methylation levels are altered in nasal epithelial and blood cell samples from CF patients. This study disclosed slightly, but significantly differentially methylated regions that collectively may modulate lung disease severity. It also highlighted that complex relationships between genetic and epigenetic factors contribute to the phenotypic variability of CF patients.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* homozygous for the F508del mutation

Exclusion Criteria:

* subjects who have an active CF exacerbation or a recent viral infection on the day of biological samples collection;
* pregnant women;
* patients who are included in interventional medical trials;
* patients who had lung transplantation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
DNA methylation levels (chemical changes) | D0 (day of inclusion)
  DNA methylation levels (chemical changes)

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël CHIRON, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UHMontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Magalhaes M, Tost J, Pineau F, Rivals I, Busato F, Alary N, Mely L, Leroy S, Murris M, Caimmi D, Claustres M, Chiron R, De Sario A. Dynamic changes of DNA methylation and lung disease in cystic fibrosis: lessons from a monogenic disease. Epigenomics. 2018 Aug;10(8):1131-1145. doi: 10.2217/epi-2018-0005. Epub 2018 Jul 27. PMID 30052057